CLINICAL TRIAL: NCT01357239
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy and Safety of AFQ056 in Adolescent Patients With Fragile X Syndrome
Brief Title: Safety and Efficacy of AFQ056 in Adolescent Patients With Fragile X Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAFQ056B2214; 2010-022638-96 (EudraCT Number)
Record Dates: First submitted 2011-05-18; First posted 2011-05-20 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Fragile X Syndrome
Keywords: Fragile X Syndrome; Martin-Bell Syndrome; Genetic Diseases; X-Linked; Escalante's syndrome
MeSH Terms: conditions — Fragile X Syndrome; Genetic Diseases, Inborn | interventions — mavoglurant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 25 mg bid (Experimental)
  Interventions: Drug: AFQ056
- 50 mg bid (Experimental)
  Interventions: Drug: AFQ056
- 100 mg bid (Experimental)
  Interventions: Drug: AFQ056
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AFQ056
  Arms: 100 mg bid; 25 mg bid; 50 mg bid
Drug: Placebo
  Arms: Placebo

SUMMARY:
This Phase IIb study is designed to assess whether 3 doses of AFQ056 are safe and effective in treating the behavioral symptoms of Fragile X Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Fragile X Syndrome, who are at least moderately ill based on a Clinical Global Impression Severity score of at least 4 and have qualifying scores on the ABC-C and IQ test at Visit 1

Exclusion Criteria:

* Advanced, severe or unstable disease that may interfere with the study outcome evaluations
* Cancer within the past 5 years, other than localized skin cancer
* Current treatment with more than two psychoactive medications, excluding anti-epileptics
* History of severe self-injurious behavior
* Weigh less than 32 kg
* Females who are sexually active

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 139 (Actual)
Dates: Start 2011-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (37):
- United States (8):
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, Decatur, Georgia
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Staten Island, New York
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Houston, Texas
- Australia (2):
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Parkville, Victoria
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
- Canada (3):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Glostrup Municipality, Denmark
- France (2):
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Paris
- Germany (5):
  - Novartis Investigative Site, Mainz, Germany
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Würzburg
- Novartis Investigative Site, Semarang, Central Java, Indonesia
- Novartis Investigative Site, Ramat Gan, Israel
- Italy (3):
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Padua
- Novartis Investigative Site, Rotterdam, Netherlands
- Spain (3):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Sant Cugat del Vallès, Catalonia
- Novartis Investigative Site, Spånga, Sweden
- Switzerland (2):
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Zurich
- Novartis Investigative Site, Istanbul, Turkey (Türkiye)
- Novartis Investigative Site, Edinburgh, United Kingdom

REFERENCES:
- [Derived] Bailey DB Jr, Berry-Kravis E, Wheeler A, Raspa M, Merrien F, Ricart J, Koumaras B, Rosenkranz G, Tomlinson M, von Raison F, Apostol G. Mavoglurant in adolescents with fragile X syndrome: analysis of Clinical Global Impression-Improvement source data from a double-blind therapeutic study followed by an open-label, long-term extension study. J Neurodev Disord. 2016;8:1. doi: 10.1186/s11689-015-9134-5. Epub 2015 Dec 15. PMID 26855682
- [Derived] Berry-Kravis E, Des Portes V, Hagerman R, Jacquemont S, Charles P, Visootsak J, Brinkman M, Rerat K, Koumaras B, Zhu L, Barth GM, Jaecklin T, Apostol G, von Raison F. Mavoglurant in fragile X syndrome: Results of two randomized, double-blind, placebo-controlled trials. Sci Transl Med. 2016 Jan 13;8(321):321ra5. doi: 10.1126/scitranslmed.aab4109. PMID 26764156

RESULTS

PARTICIPANT FLOW:
Groups:
- AFQ056 25 mg Bid: 1 capsule of 25 mg and 1 capsule of placebo per intake
- AFQ056 50 mg Bid: 2 capsules of 25 mg per intake
- AFQ056 100 mg Bid: 1 capsule of 100 mg and 1 capsule of placebo per intake
- Placebo: 2 capsules of placebo per intake
Period: Stratum: All Patients
Arm/Group | AFQ056 25 mg Bid | AFQ056 50 mg Bid | AFQ056 100 mg Bid | Placebo
Started | 31 | 27 | 39 | 42
Completed | 31 | 27 | 37 | 40
Not Completed | 0 | 0 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Subject withdrew consent | 0 | 0 | 1 | 1
Period: Stratum I: Fully-Methylated
Arm/Group | AFQ056 25 mg Bid | AFQ056 50 mg Bid | AFQ056 100 mg Bid | Placebo
Started | 8 | 6 | 17 | 22
Completed | 8 | 6 | 16 | 22
Not Completed | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Period: Stratum II: Partially-Methylated
Arm/Group | AFQ056 25 mg Bid | AFQ056 50 mg Bid | AFQ056 100 mg Bid | Placebo
Started | 23 | 21 | 22 | 20
Completed | 23 | 21 | 21 | 18
Not Completed | 0 | 0 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Subject withdrew consent | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AFQ056 25 mg Bid | AFQ056 50 mg Bid | AFQ056 100 mg Bid | Placebo | Total
Number analyzed (Participants) | 31 | 27 | 39 | 42 | 139
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.4 (1.70) | 14.6 (1.58) | 14.6 (1.77) | 14.4 (1.85) | 14.5 (1.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 4 | 3 | 15
  Male | 26 | 24 | 35 | 39 | 124

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Behavioral Symptoms of Fragile X Syndrome Using the Aberrant Behavior Checklist-Community Edition (ABC-CFX) Total Score in Stratum I Patients Exposed to AFQ056 100 mg Bid
Description: The Aberrant Behavior Checklist-Community edition (ABC-C) is a 58-item, caregiver-rated symptom checklist for assessing problem behaviors of children and adults with mental retardation at home, in residential facilities, and work training centers. The assessment was done by attributing to each item a score from 0 ("not at all a problem") to 3 ("problem is severe in degree") and the total score ranks from 0 to 174. The data collected from the full, 58-item ABC-C were analyzed according to the modified FXS ABC-C algorithm (ABC-CFX) for which 55 items and six subscales (irritability, lethargy/withdrawal, stereotypic behavior, hyperactivity, inappropriate speech and social avoidance) plus the total score were considered, and for which the total score ranks from 0 to 165. Stratum I included patients whose Fragile X Mental Retardation 1 (FMR1) gene was fully methylated
Time Frame: Baseline to week 12
Population: Full Analysis Set (FAS):all randomized patients who received at least 1 dose of study drug, had a baseline and at least 1 post-baseline assessment for the primary efficacy parameter. Only participants who had a value at the given time and the assessment was within the window for analysis were included
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | AFQ056 100 mg Bid | Placebo
Number analyzed (Participants) | 16 | 22
Score | 8.6 (4.48) | -9.4 (3.88)

2. Secondary Outcome: Change From Baseline in Behavioral Symptoms of Fragile X Syndrome Using the ABC-CFX Total Score in Stratum II Patients Exposed to All 3 Doses of AFQ056
Description: The ABC-C is a 58-item, caregiver-rated symptom checklist for assessing problem behaviors of children and adults with mental retardation at home, in residential facilities, and work training centers. The assessment was done by attributing to each item a score from 0 ("not at all a problem") to 3 ("problem is severe in degree") and the total score ranks from 0 to 174. The data collected from the full, 58-item ABC-C were analyzed according to the modified FXS ABC-C algorithm (ABC-CFX) for which 55 items and six subscales (irritability, lethargy/withdrawal, stereotypic behavior, hyperactivity, inappropriate speech and social avoidance) plus the total score were considered, and for which the total score ranks from 0 to 165. Stratum II included patients whose FMR1 gene was partially methylated
Time Frame: Baseline to week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | AFQ056 25 mg Bid | AFQ056 50 mg Bid | AFQ056 100 mg Bid | Placebo
Number analyzed (Participants) | 23 | 21 | 20 | 18
Score | -6.8 (3.88) | -2.8 (4.07) | -5.7 (4.06) | -3.5 (4.30)

3. Secondary Outcome: Change From Baseline in Behavioral Symptoms of Fragile X Syndrome Using the ABC-CFX Total Score in Stratum I Patients Exposed to the Two Lower Doses of AFQ056 (25 mg Bid and 50 mg Bid)
Description: The ABC-C is a 58-item, caregiver-rated symptom checklist for assessing problem behaviors of children and adults with mental retardation at home, in residential facilities, and work training centers. The assessment was done by attributing to each item a score from 0 ("not at all a problem") to 3 ("problem is severe in degree") and the total score ranks from 0 to 174. The data collected from the full, 58-item ABC-C were analyzed according to the modified FXS ABC-C algorithm (ABC-CFX) for which 55 items and six subscales (irritability, lethargy/withdrawal, stereotypic behavior, hyperactivity, inappropriate speech and social avoidance) plus the total score were considered, and for which the total score ranks from 0 to 165. Stratum I included patients whose FMR1 gene was fully methylated
Time Frame: Baseline to week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | AFQ056 25 mg Bid | AFQ056 50 mg Bid | Placebo
Number analyzed (Participants) | 8 | 6 | 22
Score | -11.8 (6.43) | -3.4 (7.40) | -9.4 (3.88)

4. Secondary Outcome: Global Improvement of Symptoms in Fragile X Using the Clinical Global Impression- Improvement (CGI-I) Scale in Stratum I Patients
Description: The Clinical Global Impression-Improvement (CGI-I) scale is a clinician rated scale used to assess treatment response in psychiatric patients, and the score ranges from 1 to 7 (with 1 being "very much improved", 4 being "no change" to 7 being "very much worse"). Stratum I included patients whose FMR1 gene was fully methylated.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | AFQ056 25 mg Bid | AFQ056 50 mg Bid | AFQ056 100 mg Bid | Placebo
Number analyzed (Participants) | 8 | 6 | 15 | 22
Score | 3.3 (0.30) | 3.8 (0.34) | 3.5 (0.22) | 3.1 (0.18)

5. Secondary Outcome: Global Improvement of Symptoms in Fragile X Using the Clinical Global Impression- Improvement (CGI-I) Scale in Stratum II Patients
Description: The Clinical Global Impression-Improvement (CGI-I) scale is a clinician rated scale used to assess treatment response in psychiatric patients, and the score ranges from 1 to 7 (with 1 being "very much improved", 4 being "no change" to 7 being "very much worse"). Stratum II included patients whose FMR1 gene was partially methylated
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | AFQ056 25 mg Bid | AFQ056 50 mg Bid | AFQ056 100 mg Bid | Placebo
Number analyzed (Participants) | 23 | 21 | 20 | 18
Score | 3.5 (0.19) | 3.2 (0.20) | 3.5 (0.20) | 3.4 (0.21)

6. Secondary Outcome: Global Improvement of Symptoms in Fragile X Using the Clinical Global Impression-Improvement (CGI-I) Scale in Stratum I
Description: as for outcome 4
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | AFQ056 25 mg Bid | AFQ056 50 mg Bid | AFQ056 100 mg Bid | Placebo
Number analyzed (Participants) | 8 | 6 | 15 | 22
Participants
  1 (Very much improved) | 1 (0.30) | 0 (0.34) | 0 (0.22) | 0 (0.18)
  2 (Much improved) | 0 (0.19) | 0 (0.20) | 3 (0.20) | 4 (0.21)
  3 (Minimally improved) | 2 | 1 | 3 | 11
  4 (No change) | 5 | 5 | 6 | 6
  5 (Minimally worse) | 0 | 0 | 3 | 1
  6 (Much worse) | 0 | 0 | 0 | 0
  7 (Very much worse) | 0 | 0 | 0 | 0

7. Secondary Outcome: Global Improvement of Symptoms in Fragile X Using the Clinical Global Impression-Improvement (CGI-I) Scale in Stratum II
Description: as for outcome 5
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | AFQ056 25 mg Bid | AFQ056 50 mg Bid | AFQ056 100 mg Bid | Placebo
Number analyzed (Participants) | 23 | 21 | 20 | 18
Participants
  1 (Very much improved) | 0 (0.30) | 0 (0.34) | 0 (0.22) | 0 (0.18)
  2 (Much improved) | 3 (0.19) | 5 (0.20) | 3 (0.20) | 4 (0.21)
  3 (Minimally improved) | 7 | 9 | 4 | 5
  4 (No change) | 12 | 5 | 11 | 8
  5 (Minimally worse) | 1 | 2 | 2 | 0
  6 (Much worse) | 0 | 0 | 0 | 1
  7 (Very much worse) | 0 | 0 | 0 | 0

8. Secondary Outcome: Change From Baseline in Irritability, Lethargy/Withdrawal, Stereotypic Behavior, Hyperactivity, Inappropriate Speech and Social Avoidance Assessed by the Individual Subscales of the ABC-CFX Scale in Stratum I
Description: The ABC-C is a 58-item, caregiver-rated symptom checklist for assessing problem behaviors of children and adults with mental retardation at home, in residential facilities, and work training centers. The assessment was done by attributing to each item a score from 0 ("not at all a problem") to 3 ("problem is severe in degree") and the total score ranks from 0 to 174. The data collected from the full, 58-item ABC-C were analyzed according to the modified FXS ABC-C algorithm (ABC-CFX) for which 55 items and six subscales: irritability (range 0 to 54); lethargy/withdrawal (range 0 to 39); stereotypic behavior (range 0 to 18); hyperactivity (range 0 to 30); inappropriate speech (range 0 to 12); and social avoidance (range 0 to 12) plus the total score (range 0 to 165) were considered. A negative change represents improvement. Stratum I included patients whose FMR1 gene was fully methylated
Time Frame: Baseline to week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | AFQ056 25 mg Bid | AFQ056 50 mg Bid | AFQ056 100 mg Bid | Placebo
Number analyzed (Participants) | 8 | 6 | 16 | 22
Score
  Irritability | -3.5 (2.74) | 2.2 (3.21) | 4.2 (1.94) | -2.5 (1.67)
  Lethargy/withdrawal | -1.4 (1.29) | -3.5 (1.53) | 1.3 (0.92) | -1.9 (0.78)
  Stereotypic behavior | -2.2 (0.96) | -2.2 (1.10) | 1.2 (0.67) | -1.7 (0.58)
  Hyperactivity | -3.9 (1.57) | 1.1 (1.78) | 0.7 (1.09) | -1.3 (0.95)
  Inappropriate speech | -0.8 (0.69) | 0.3 (0.78) | 0.9 (0.48) | -1.0 (0.42)
  Social avoidance | -0.2 (0.71) | -1.0 (0.80) | -0.1 (0.50) | -1.2 (0.42)

9. Secondary Outcome: Change From Baseline in Irritability, Lethargy/Withdrawal, Stereotypic Behavior, Hyperactivity, Inappropriate Speech, and Social Avoidance Assessed by the Individual Subscales of the ABC-CFX Scale in Stratum II
Description: The ABC-C is a 58-item, caregiver-rated symptom checklist for assessing problem behaviors of children and adults with mental retardation at home, in residential facilities, and work training centers. The assessment was done by attributing to each item a score from 0 ("not at all a problem") to 3 ("problem is severe in degree") and the total score ranks from 0 to 174. The data collected from the full, 58-item ABC-C were analyzed according to the modified FXS ABC-C algorithm (ABC-CFX) for which 55 items and six subscales: irritability (range 0 to 54); lethargy/withdrawal (range 0 to 39); stereotypic behavior (range 0 to 18); hyperactivity (range 0 to 30); inappropriate speech (range 0 to 12); and social avoidance (range 0 to 12) plus the total score (range 0 to 165) were considered. A negative change represents improvement. Stratum II included patients whose FMR1 gene was partially methylated
Time Frame: Baseline to week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | AFQ056 25 mg Bid | AFQ056 50 mg Bid | AFQ056 100 mg Bid | Placebo
Number analyzed (Participants) | 23 | 21 | 20 | 18
Score
  Irritability | -1.5 (1.58) | -1.3 (1.65) | -0.8 (1.66) | 0.0 (1.75)
  Lethargy/withdrawal | -0.8 (1.00) | -0.4 (1.05) | -0.3 (1.05) | -0.8 (1.11)
  Stereotypic behavior | -1.4 (0.57) | 0.1 (0.60) | -1.0 (0.60) | 0.1 (0.64)
  Hyperactivity | -1.5 (0.87) | -0.3 (0.91) | -1.8 (0.91) | -0.8 (0.96)
  Inappropriate speech | -0.9 (0.44) | -0.1 (0.46) | -0.6 (0.47) | -0.8 (0.50)
  Social avoidance | -0.7 (0.40) | -0.9 (0.42) | -1.1 (0.42) | -1.1 (0.45)

10. Secondary Outcome: Proportion of Patients With Clinical Response, Where Response is Defined as a Reduction of at Least 25% From Baseline in the ABC-CFX Total Score and a Score of 1 (Very Much Improved) or 2 (Much Improved) on the CGI-I Scale, Stratum I
Description: The ABC-C is a 58-item, caregiver-rated symptom checklist for assessing problem behaviors of children and adults with mental retardation at home, in residential facilities, and work training centers. The assessment was done by attributing to each item a score from 0 ("not at all a problem") to 3 ("problem is severe in degree") and the total score ranks from 0 to 174. The data collected from the full, 58-item ABC-C were analyzed according to ABC-CFX algorithm, for which 55 items and six subscales plus the total score were considered, and for which the total score ranks from 0 to 165. The Clinical Global Impression-Improvement (CGI-I) scale is a clinician rated scale used to assess treatment response in psychiatric patients, and the score ranges from 1 to 7 (with 1 being "very much improved", 4 being "no change" to 7 being "very much worse"). Stratum I included patients whose FMR1 gene was fully methylated; Stratum II included patients whose FMR1 gene was partially methylated.
Time Frame: 12 weeks
Population: Full Analysis Set (FAS):all randomized patients who received at least 1 dose of study drug, had a baseline and at least 1 post-baseline assessment for the primary efficacy parameter. Total is the number of patients with non-missing baseline ABC-CFX total score and at least one nonmissing post-baseline ABC-CFX total score and CGI-I assessment
Measure: Number; unit: Number of participants
Arm/Group | AFQ056 25 mg Bid | AFQ056 50 mg Bid | AFQ056 100 mg Bid | Placebo
Number analyzed (Participants) | 8 | 6 | 17 | 22
Number of participants | 1 | 0 | 1 | 2

11. Secondary Outcome: Proportion of Patients With Clinical Response, Where Response is Defined as a Reduction of at Least 25% From Baseline in the ABC-CFX Total Score and a Score of 1 (Very Much Improved) or 2 (Much Improved) on the CGI-I Scale, Stratum II
Description: as for outcome 10
Time Frame: 12 weeks
Population: as for outcome 10
Measure: Number; unit: Number of participants
Arm/Group | AFQ056 25 mg Bid | AFQ056 50 mg Bid | AFQ056 100 mg Bid | Placebo
Number analyzed (Participants) | 23 | 21 | 22 | 19
Number of participants | 1 | 4 | 1 | 2

12. Secondary Outcome: Change From Baseline in Repetitive Behaviors Assessed Using the Repetitive Behavior Scale - Revised (RBS-R) Total and Subscale Scores in Stratum I
Description: The Repetitive Behavior Scale - Revised (RBS-R) is a rating tool that captures the breadth of repetitive behavior. It is a 43-item questionnaire filled by the caregivers. Each behavior assessed is rated from 0 (behavior does not occur) to 3 (behavior occurs and it is a severe problem). The total score ranks from 0 to 129. The behaviors are grouped into six domains: ritualistic behavior (range 0 to 18); sameness behavior (range 0 to 33); stereotypic behavior (range 0 to 18); self-injurious behavior (range 0 to 24); compulsive behavior (range 0 to 24); and restricted interests (range 0 to 12). A negative change represents improvement. Stratum I included patients whose FMR1 gene was fully methylated
Time Frame: Baseline to week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | AFQ056 25 mg Bid | AFQ056 50 mg Bid | AFQ056 100 mg Bid | Placebo
Number analyzed (Participants) | 8 | 6 | 16 | 22
Score on a scale
  Total score | -2.3 (3.25) | -8.5 (3.95) | 1.5 (2.31) | -6.2 (2.03)
  Stereotyped behavior | -1.0 (0.91) | -1.5 (1.03) | 0.5 (0.64) | -1.0 (0.56)
  Self-injurious behavior | 0.0 (0.46) | 0.8 (0.53) | -0.2 (0.33) | -1.1 (0.28)
  Compulsive behavior | -0.1 (0.84) | -1.2 (1.06) | 0.2 (0.60) | -0.8 (0.51)
  Ritualistic behavior | -0.2 (0.93) | -2.2 (1.12) | 0.8 (0.66) | -0.6 (0.57)
  Sameness behavior | -0.8 (1.19) | -2.8 (1.42) | 0.3 (0.85) | -1.8 (0.73)
  Restricted behavior | 0.0 (0.65) | -1.2 (0.74) | -0.2 (0.46) | -1.1 (0.39)

13. Secondary Outcome: Change From Baseline in Repetitive Behaviors Assessed Using the Repetitive Behavior Scale - Revised (RBS-R) Total and Subscale Scores in Stratum II
Description: The Repetitive Behavior Scale - Revised (RBS-R) is a rating tool that captures the breadth of repetitive behavior. It is a 43-item questionnaire filled by the caregivers. Each behavior assessed is rated from 0 (behavior does not occur) to 3 (behavior occurs and it is a severe problem). The total score ranks from 0 to 129. The behaviors are grouped into six domains: ritualistic behavior (range 0 to 18); sameness behavior (range 0 to 33); stereotypic behavior (range 0 to 18); self-injurious behavior (range 0 to 24); compulsive behavior (range 0 to 24); and restricted interests (range 0 to 12). A negative change represents improvement. Stratum II included patients whose FMR1 gene was partially methylated
Time Frame: Baseline to week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | AFQ056 25 mg Bid | AFQ056 50 mg Bid | AFQ056 100 mg Bid | Placebo
Number analyzed (Participants) | 23 | 21 | 20 | 18
Score on a scale
  Total score | -4.3 (2.36) | -5.9 (2.51) | -2.4 (2.47) | -5.0 (2.67)
  Stereotyped behavior | 0.1 (0.53) | 0.1 (0.56) | 0.4 (0.56) | 0.2 (0.59)
  Self-injurious behavior | -0.6 (0.53) | -0.7 (0.55) | 0.0 (0.56) | 0.5 (0.59)
  Compulsive behavior | -0.9 (0.58) | -1.5 (0.62) | -0.2 (0.61) | -1.0 (0.65)
  Ritualistic behavior | -0.1 (0.55) | -1.5 (0.58) | -1.0 (0.58) | -1.8 (0.62)
  Sameness behavior | -2.2 (0.77) | -1.6 (0.83) | -1.3 (0.82) | -2.8 (0.88)
  Restricted behavior | -0.6 (0.40) | -0.7 (0.43) | -0.4 (0.42) | -0.3 (0.45)

ADVERSE EVENTS:
Arm/Group | Placebo | AFQ056 25 mg Bid | AFQ056 50 mg Bid | AFQ056 100 mg Bid
Serious Adverse Events (participants affected / at risk) | 2/42 | 0/31 | 0/27 | 0/39
Other Adverse Events (participants affected / at risk) | 17/42 | 22/31 | 9/27 | 30/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=42) | AFQ056 25 mg Bid (N=31) | AFQ056 50 mg Bid (N=27) | AFQ056 100 mg Bid (N=39)
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=42) | AFQ056 25 mg Bid (N=31) | AFQ056 50 mg Bid (N=27) | AFQ056 100 mg Bid (N=39)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1 | 6
Fatigue (General disorders) | 0 | 0 | 1 | 2
Pyrexia (General disorders) | 1 | 2 | 1 | 3
Influenza (Infections and infestations) | 2 | 2 | 0 | 2
Nasopharyngitis (Infections and infestations) | 6 | 7 | 6 | 5
Oral herpes (Infections and infestations) | 0 | 2 | 0 | 2
Rhinitis (Infections and infestations) | 0 | 2 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 2 | 1 | 5
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 4
Headache (Nervous system disorders) | 4 | 4 | 0 | 10
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 2
Initial insomnia (Psychiatric disorders) | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 6
Self injurious behaviour (Psychiatric disorders) | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety